CLINICAL TRIAL: NCT00778518
Title: Phase IIb Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profile of ARX201 Following Repeated Dosing to Young Adult Patients With Childhood Onset Growth Hormone Deficiency (GHD).
Brief Title: Safety, Tolerability and PK/PD Study in Young Adult Patients With Childhood Onset Growth Hormone Deficiency (GHD).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ambrx, Inc. (Industry)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Douglas W. Axelrod, MD, PhD, Sr. Vice President, Clinical Research and Development, Ambrx, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-ARX201-701; EudraCT: 2007-001746-40
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Growth Hormone Deficiency
Keywords: growth hormone; growth hormone deficiency; GHD; PEG; pegylated; IGF-1
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): low dose
  Interventions: Drug: ARX201
- 2 (Active Comparator): Medium dose
  Interventions: Drug: ARX201
- 3 (Active Comparator): High Dose
  Interventions: Drug: ARX201

INTERVENTIONS:
Drug: ARX201 — Reconstituted lyophilized drug product at 2.5 mg/wk; 3 periods over six months.
  Arms: 1
Drug: ARX201 — Reconstituted lyophilized drug product at 5.0 mg/wk; 3 periods over six months.
  Arms: 2
Drug: ARX201 — Reconstituted lyophilized drug product at 10.0 mg/wk; 3 periods over six months.
  Arms: 3

SUMMARY:
Study to find the optimal dose of Growth Hormone Replacement in young adult patients suffering from childhood onset growth hormone deficiency (GHD).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety, tolerability and pharmacodynamic response of three different ARX201 doses (PEG-ahGH) when administered repeatedly to young adult patients with childhood onset growth hormone deficiency (GHD).

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* GHD of childhood onset
* completed growth
* IGF-1 <=2SDS
* rhGH treatment naive
* hGH levels below cut-off

Exclusion Criteria:

* History of malignancy or intracranial tumors
* ECG abnormality
* ICH
* hepatic dysfunction
* renal impairment
* major medical conditions
* inadequate T4
* positive for HBV, HCV, or HIV
* alcohol or drug abuse

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Temporal profiling of circulating IGF-1 levels. | 3 period

SECONDARY OUTCOMES:
Body composition measurements at start of study and end of study | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mihaly Juhasz, MD, Study Director — Accelsiors CRO & Consultancy Services
Locations (1):
- Accelsiors CRO and Consultancy Services, Budapest, Hungary